CLINICAL TRIAL: NCT05913726
Title: Network of Doctors for Multimorbidity and Diabetes - The NOMAD Intervention: Protocol for Feasibility Trial of Multidisciplinary Team Conferences for People With Diabetes and Multimorbidity
Brief Title: MDT Conferences for People With Diabetes and Multimorbidity
Acronym: NOMAD
Status: Completed | Type: Observational
Sponsor: Odense University Hospital (Other)
Collaborators: Steno Diabetes Center Odense (Other)
Responsible Party: Principal Investigator, Stine Jorstad Bugge, Ph.d. student and MD, Odense University Hospital
Other Study IDs: Steno-MDT3
Record Dates: First submitted 2023-04-26; First posted 2023-06-22 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Diabetes Mellitus; Comorbidities and Coexisting Conditions
Keywords: Multidisciplinary team conferences; Feasibility
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to test if regular meetings (multidisciplinary team conferences) between several different medical doctors can work well in everyday hospital life. The doctor meetings are meant to discuss patients who have both diabetes and other chronic conditions at the same time.

The main questions it aims to answer are:

* How can the concept of these meetings work in everyday hospital life?
* What are the patients and doctors getting out of the meetings?

Patients with diabetes and concurrent other diseases will be asked:

* if they want their case discussed on the doctor meeting
* to answer a set of questions about their well-being and symptoms before and 6 months after the meeting
* if the research group can store their information for the study

Doctors participating in the meetings are asked to answer questions about what they have learned in the meetings.

DETAILED DESCRIPTION:
Introduction: Many people struggle with several chronic conditions at once. This is known as multimorbidity. The prevalence of multimorbidity is rising. Diabetes is one of the chronic conditions often associated with multimorbidity. The prevalence of diabetes is likewise increasing world-wide.

Having diabetes and multimorbidity can be a great burden for a person as they have to deal with symptoms, treatments, lifestyle changes and checkups. The picture complicates as many healthcare systems have a disease-specific approach rather than a patient-centered approach. This often leads to multiple different outpatient clinic contacts, possibly uncoordinated treatment and fragmented care. One can view the patient as a nomad between departments and sectors, often lacking coherence.

The aim of this study is to feasibility test a complex intervention designed to coordinate care and treatment for people with diabetes and multimorbidity prior to a large-scale randomised trial.

Intervention: To gain a more patient-centered approach, better coordination of care and treatment and possibly increase life quality for people with diabetes and multimorbidity, a working group has set out to develop a complex intervention guided by relevant guidelines. The intervention consists of multidisciplinary team conferences (MDT) performed by medical doctors within the specialities of endocrinology, cardiology, respiratory medicine, nephrology and clinical pharmacology, called Network of dOctors for Multimorbidity and Diabetes - NOMAD. The doctors sit together every two weeks to discuss the treatment, coordinate care and review medications of referred patients with diabetes and minimum one other condition within the collaborating specialities. Patients can be referred from hospital departments or from their general practitioner (GP), in which case, the GP attends the meeting by video conference. Prior to the MDT, a questionnaire concerning health related quality of life is sent out to the patient. The same questionnaire is sent out 6 months after the MDT and followed by a contact to the patient - either physical or by phone by healthcare professional. The doctors review the answers before the MDT and use them as discussion support in the MDT. All doctors attending the MDT have time scheduled prior to MDT to prepare and read about the patients. Especially the clinical pharmacologist has extended preparation time to ensure a thorough review of the patients medications list - which oftentimes consist of more than 15 different prescriptions.

Methods: This is a one-arm mixed-methods feasibility study of a complex intervention. The MDT conferences will be evaluated for feasibility through prospectively collected data. The evaluation will be based on the following process indicators:

1. completion of PRO-questionnaire
2. technical issues before, during or after MDT
3. time schedule in MDT kept or not
4. does MDT conclusion note correspond to MDT referral letter?
5. clinician preparation time

The patients' perspectives will be explored through the questionnaires and also through interviews of a selection of participants - both intervention receivers and providers, contributing to a qualitative process evaluation. The feasibility of using (patient-reported outcome, PRO) a collection of generic, validated questionnaires to measure intervention effect will be assessed. Through a run-time of 17 months, approximately 120 participants are anticipated. Results will be reported narratively and with descriptive statistics. The interviews will be reported in a separate paper.

Ethics: As the study focuses mainly on an organisational level, detailed information on individual level is not required. The scientific ethics committee has been requested for approval, replying that this study is exempt from ethics approval as it collects no human material (ref. number: 20222000 - 150).

The study is registered in list of research/quality-development projects in Region of Southern Denmark (ref. number: 22/56265).

Implications: This study will provide valuable insights into how a complex intervention of MDTs can be implemented in clinical practice, how it is received by end-users and provide decision-makers with useful experience on how to organise such an intervention. Furthermore it will elucidate the use of PRO and laboratory values as effect measures. All of this will lay the grounds for a future randomised trial where efficiency, effectiveness and clinical effect of MDT can be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Adult, any type of diabetes, diabetes management by general practitioner or Steno Diabetes Centre Odense, minimum one chronic condition within heart, kidney or lung specialities.

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study population consists of all adult residents in the geographical region of Funen, Denmark, who meet eligibility criteria.
  Funen inhabits approximately 500.000.
Sampling Method: Non-Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-07-01 (Actual)

PRIMARY OUTCOMES:
Recruitment | Full project period, 17 months.
  Number of patients referred to MDT. Reported as total number of referred patients throughout the project period and as mean/median per MDT.
Completion of PRO-questionnaire | Full project period, 17 months.
  How many participants completed the PRO-questionnaire. Reported as absolute number and percentage of total number of participants.
Technical difficulties i relation to MDT | Full project period, 17 months.
  How many times did technical difficulties occur i relation to MDT. Technical difficulties defined as 1) problem with sending/receiving referral letter, 2) managing PRO-questionnaire completion, 3) problems with video, sound or connection during MDT or 4) problems with contacting participant for followup. Reported as absolute numbers and percentage of all MDTs.
Time schedule | Full project period, 17 months.
  Was time schedule kept on MDT? Simple count of how often time schedule of 30 minutes per patient case was NOT kept. Reported as absolute number and percentage of total number of patient cases.
MDT recommendations | Assessed at 6 month follow up.
  How often are MDT recommendations initiated? Assessed at 6 month follow up by examining electronic patient records and conversation with participant. Reported as simple count of how many times recommendations are followed/initiated and percentage of recommendations followed out of total MDT recommendations.
Clinician preparation time | Full project period, 17 months.
  How many minutes does each clinician take to prepare an MDT case discussion? Assessed by survey completed by clinicians at end of each MDT case discussion. Reported as means and medians in whole minutes.

SECONDARY OUTCOMES:
Laboratory values | Assessed at time point of referral to MDT and 6 months after MDT.
  A simple count of how many participants who have relevant laboratory values (HbA1C, LDL, creatinine) less than 90 days old at time point of referral and time point of 6 months follow up. Reported as absolute numbers and percentages.
Clinician learning | Full project period, 17 months.
  To which degree did the clinician find the MDT case discussion educational/enlightening/useful for personal development? Assessed by completion of mini-survey by each clinician at the end of each MDT case discussion. Survey consists of visual analogue scale 0-100 mm. 0 indicating "not educational at all" and 100 indicating "most educational, as much as possible". Clinician learning is reported as means and medians on this scale.

CONTACTS AND LOCATIONS:
Overall Officials: Ann-Dorthe O Zwisler, Professor, Principal Investigator — Dept.s of Cardiology and Clinical Research, O.U. Hospital and University of Southern Denmark.
Locations (1):
- Odense University Hospital, Odense, Denmark

IPD SHARING:
Plan to Share IPD: No
The results will be published and shared in an international peer-reviewed journal.

REFERENCES:
- [Background] Uijen AA, van de Lisdonk EH. Multimorbidity in primary care: prevalence and trend over the last 20 years. Eur J Gen Pract. 2008;14 Suppl 1:28-32. doi: 10.1080/13814780802436093. PMID 18949641
- [Background] Saeedi P, Petersohn I, Salpea P, Malanda B, Karuranga S, Unwin N, Colagiuri S, Guariguata L, Motala AA, Ogurtsova K, Shaw JE, Bright D, Williams R; IDF Diabetes Atlas Committee. Global and regional diabetes prevalence estimates for 2019 and projections for 2030 and 2045: Results from the International Diabetes Federation Diabetes Atlas, 9th edition. Diabetes Res Clin Pract. 2019 Nov;157:107843. doi: 10.1016/j.diabres.2019.107843. Epub 2019 Sep 10. PMID 31518657
- [Background] Williams JS, Egede LE. The Association Between Multimorbidity and Quality of Life, Health Status and Functional Disability. Am J Med Sci. 2016 Jul;352(1):45-52. doi: 10.1016/j.amjms.2016.03.004. Epub 2016 Mar 18. PMID 27432034
- [Background] Skivington K, Matthews L, Simpson SA, Craig P, Baird J, Blazeby JM, Boyd KA, Craig N, French DP, McIntosh E, Petticrew M, Rycroft-Malone J, White M, Moore L. A new framework for developing and evaluating complex interventions: update of Medical Research Council guidance. BMJ. 2021 Sep 30;374:n2061. doi: 10.1136/bmj.n2061. PMID 34593508
- [Background] O'Cathain A, Croot L, Duncan E, Rousseau N, Sworn K, Turner KM, Yardley L, Hoddinott P. Guidance on how to develop complex interventions to improve health and healthcare. BMJ Open. 2019 Aug 15;9(8):e029954. doi: 10.1136/bmjopen-2019-029954. PMID 31420394
- [Background] Henriksen DP, Ennis ZN, Panou V, Hangaard J, Jensen PB, Johansson SL, Nagarajah S, Poulsen MK, Rothmann MJ, Schousboe K, Bugge SJ, Jessen LB, Schneider IR, Olsen Zwisler AD, Hojlund K, Damkier P. Physician-led in-hospital multidisciplinary team conferences with multiple medical specialities present - A scoping review. J Multimorb Comorb. 2022 Dec 7;12:26335565221141745. doi: 10.1177/26335565221141745. eCollection 2022 Jan-Dec. PMID 36518524
- [Background] Andersen JD, Jensen MH, Vestergaard P, Jensen V, Hejlesen O, Hangaard S. The multidisciplinary team in diagnosing and treatment of patients with diabetes and comorbidities: A scoping review. J Multimorb Comorb. 2023 Mar 20;13:26335565231165966. doi: 10.1177/26335565231165966. eCollection 2023 Jan-Dec. PMID 36968789
- [Background] Fortin M, Lapointe L, Hudon C, Vanasse A, Ntetu AL, Maltais D. Multimorbidity and quality of life in primary care: a systematic review. Health Qual Life Outcomes. 2004 Sep 20;2:51. doi: 10.1186/1477-7525-2-51. PMID 15380021
- [Background] Menotti A, Mulder I, Nissinen A, Giampaoli S, Feskens EJ, Kromhout D. Prevalence of morbidity and multimorbidity in elderly male populations and their impact on 10-year all-cause mortality: The FINE study (Finland, Italy, Netherlands, Elderly). J Clin Epidemiol. 2001 Jul;54(7):680-6. doi: 10.1016/s0895-4356(00)00368-1. PMID 11438408
- [Derived] Bugge SJ, Henriksen DP, Damkier P, Rahbek MT, Schousboe K, Rothmann MJ, Poulsen MK, Hansen C, Nagarajah S, Jensen PB, Johansson SL, Panou V, Schneider IR, Pedersen CG, Andersen JD, Hangaard J, Zwisler AO. Network of doctors for multimorbidity and diabetes - the NOMAD intervention: protocol for feasibility trial of multidisciplinary team conferences for people with diabetes and multimorbidity. Pilot Feasibility Stud. 2024 Jun 15;10(1):91. doi: 10.1186/s40814-024-01517-0. PMID 38879561
- See also: World Health Organization. Multimorbidity. Geneva. ; 2016. ISBN 978-92-4-151165-0 — https://apps.who.int/iris/bitstream/handle/10665/252275/9789241511650-eng.pdf
- See also: Invisible numbers: the true extent of noncommunicable diseases and what to do about them. Geneva: World Health Organization; 2022. Licence: CC BY-NC-SA 3.0 IGO. — https://www.who.int/publications/i/item/9789240057661